CLINICAL TRIAL: NCT03485001
Title: Treatment of Primary Type I Pterygia With Argon Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CC-08-2011
Record Dates: First submitted 2016-12-28; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Sham of Argon Laser Treatment (Sham Comparator): Slit lamp light exposure
  Interventions: Other: Sham
- Argon Laser Treatment (Experimental): Argon Laser Treatment
  Interventions: Procedure: Argon Laser Treatment

INTERVENTIONS:
Other: Sham — This group will not receive argon laser medical treatment; instead, they will be only exposed to the slit lamp light.
  Arms: Sham of Argon Laser Treatment
Procedure: Argon Laser Treatment — This group will receive argon laser medical treatment to the body and head of pterygium
  Arms: Argon Laser Treatment

SUMMARY:
Introduction: Pterygium is a wing shape degenerative and hyperplastic growth of the bulbar conjunctiva extending onto the cornea, most commonly on the nasal side. Management of pterygium can be medical, surgical or combined. Alternative treatments as photocoagulation of blood vessels of the pterygium, have been described, especially in recurrent pterygia.

Objectives: To determine whether Argon laser treatment reduces the symptoms and pterygium size in primary type I pterygia patients when compared with medical treatment. Subjects and Methods: Prospective, comparative and interventional study. Patients with type I pterygia in both eyes were included. The eyes were randomly divided to receive either Argon laser treatment or only topical medical treatment

DETAILED DESCRIPTION:
Pterygium is a wing shape degenerative and hyperplastic growth of the bulbar conjunctiva extending onto the cornea, most commonly on the nasal side. Management of pterygium can be medical, surgical or combined. Alternative treatments as photocoagulation of blood vessels of the pterygium, have been described, especially in recurrent pterygia.

To determine whether Argon laser treatment reduces the symptoms and pterygium size in primary type I pterygia patients when compared with medical treatment. Subjects and Methods: Prospective, comparative and interventional study. Patients with type I pterygia in both eyes were included. The eyes were randomly divided to receive either Argon laser treatment or only topical medical treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients who had had symmetric type I pterygia in both eyes
* Assessments for the 6 month follow-up period after argon laser treatment

Exclusion Criteria:

* Patients with diabetes Mellitus, collagenopathies, previous ocular surgeries, and pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pterygia measurements | 1 year
  Measurements were performed according to Welch et al. modified technique as following: the distance in millimeters from the limbus to the apex of the lesion on the cornea (horizontal length) was performed using the slit-lamp beam (BQ 900, Haag-Streit, Koeniz, Switzerland). A standard magnification of 16 was used and the variable aperture was focused from the limbus to the apex.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología, Mexico City, Mexico

REFERENCES:
- [Background] Welch MN, Reilly CD, Kalwerisky K, Johnson A, Waller SG. Pterygia measurements are more accurate with anterior segment optical coherence tomography - a pilot study. Nepal J Ophthalmol. 2011 Jan-Jun;3(1):9-12. doi: 10.3126/nepjoph.v3i1.4271. PMID 21505540
- [Background] Nava-Castaneda A, Tovilla-Canales JL, Rodriguez L, Tovilla Y Pomar JL, Jones CE. Effects of lacrimal occlusion with collagen and silicone plugs on patients with conjunctivitis associated with dry eye. Cornea. 2003 Jan;22(1):10-4. doi: 10.1097/00003226-200301000-00003. PMID 12502940